CLINICAL TRIAL: NCT04510935
Title: Effects of Serum From Hepatocellular Carcinoma Surgery Patients Under Different Anesthetic Methods on Hepatic Cancer Cell Function in Vitro
Brief Title: Effects of Anesthetic Methods on Hepatic Cancer Cell Function in Vitro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Jie Tian, Principle Investigator, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HCCRA202008
Record Dates: First submitted 2020-08-09; First posted 2020-08-12 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Anesthesia, General; Anesthesia, Local

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- general anesthesia (Experimental): Patients in this group will have RF ablation for treatment of HCC under general anesthesia.
  Interventions: Procedure: general anesthesia
- local anesthesia (Active Comparator): In this group, patients will receive radiofrequency ablation under local anesthesia.
  Interventions: Procedure: local anesthesia

INTERVENTIONS:
Procedure: general anesthesia — the patient will receive general anesthesia during surgery in this group.
  Arms: general anesthesia
Procedure: local anesthesia — the patient will receive local anesthesia during surgery in this group.
  Arms: local anesthesia

SUMMARY:
Numerous studies find that anesthetic methods may influence the recurrence of tumor and the overall survival of patients after primary cancer surgery. Radiofrequency (RF) ablation is now widely used in the clinic for treatment of hepatocellular carcinoma (HCC). Currently, diverse anesthetic methods, including general anesthesia (GA), epidural anesthesia and local anesthesia (LA), are used for RF ablation surgery. Using serum from HCC surgery patients randomized to receive either GA or LA during surgery, we will investigate the effects of anesthetic methods on cellular invasion, migration and proliferation of HepG2 hepatic cancer cells in vitro. The expression levels of inflammatory cytokines in the serum from patients of both groups will also be analyzed.

DETAILED DESCRIPTION:
Patients diagnosed with hepatocellular carcinoma (HCC) undergoing elective radiofrequency (RF) ablation surgery will be randomly allocated to general anesthesia(GA) group or local anesthesia(LA) group.

Patients from GA group will receive anesthesia induced with 0.05-0.1mg/kg intravenous midazolam, 3-6ug/kg fentanyl, 1.0-2.5mg/kg propofol and 0.1-0.2mg/kg atracurium. Laryngeal mask will be used to maintain ventilation. Anesthesia will be maintained with 4-8mg/kg/h propofol and 0.1-0.3ug/kg/min remifentanil, and additional non-depolarizing muscle relaxant when necessary. In patients from LA group, analgesia will be provided by a subcutaneous injection of 2% lidocaine by the surgeons before insertion of the needles.

Serum will be collected from patients of both groups at before induction and 1h post-surgery. The HepG2 hepatic cancer cell line will be treated with patient serum from both groups. The effects of anesthetic methods on cellular invasion, migration, proliferation will be measured. The expression levels of inflammatory cytokines in the serum from patients of both groups will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old
* ASA grade I-III
* Diagnosed with a single primary liver tumor of 3cm or smaller
* Is scheduled for elective radiofrequency ablation surgery
* With no macro-vascular invasion, no lymph node or extrahepatic metastases
* Child-Pugh Class A or B

Exclusion Criteria:

* a history of liver surgery previously (including radiofrequency ablation)
* severe systemic disease (heart, lung, kidney, or immune system)
* INR>1.5 or platelet count <45,000 cells/mm3
* a history of addiction to opioids;
* Disagree to participate the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-28 (Actual)

PRIMARY OUTCOMES:
mean percentage change from post- to pre-operative values of invasion of HepG2 cells cultured in patients' serum | at 1 hour post-surgery
  HepG2 cells will be cultured with serum from patients undergoing RF ablation under GA or LA for 24h. Cell invasion will be measured with Matrigel methods. Mean percentage change from post- to pre-operative values of invasion for each individual patient will be calculated and compared between the GA and LA groups.

SECONDARY OUTCOMES:
mean percentage change from post- to pre-operative values of migration of HepG2 cells cultured in patients' serum | at 1 hour post-surgery
  HepG2 cells will be cultured with serum from patients undergoing RF ablation under GA or LA for 24h. Cell migration will be measured with Transwell methods. Mean percentage change from post- to pre-operative values of migration for each individual patient will be calculated and compared between the GA and LA groups.
mean percentage change from post- to pre-operative values of proliferation of HepG2 cells cultured in patients' serum | at 1 hour post-surgery
  HepG2 cells will be cultured with serum from patients undergoing RF ablation under GA or LA for 24h. Cell proliferation will be measured with EdU methods. Mean percentage change from post- to pre-operative values of proliferation for each individual patient will be calculated and compared between the GA and LA groups.
serum IL-1β level | at 1 hour post-surgery
  an inflammatory mediator that reflects systemic inflammation
serum IL-6 level | at 1 hour post-surgery
  an inflammatory mediator that reflects systemic inflammation
serum TNF-α level | at 1 hour post-surgery
  an inflammatory mediator that reflects systemic inflammation
serum IFN-gamma level | at 1 hour post-surgery
  an inflammatory mediator that reflects systemic inflammation
serum IL-2 level | at 1 hour post-surgery
  an inflammatory mediator that reflects systemic inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Jie Tian, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital affliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided